CLINICAL TRIAL: NCT03017430
Title: Randomized Clinical Trial of Pregabalin for Opioid Withdrawal Syndrome
Brief Title: Pregabalin for Opiate Withdrawal Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Petersburg Bekhterev Research Psychoneurological Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRPI-PGBL-OW01
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Opioid Withdrawal
MeSH Terms: interventions — Pregabalin; Clonidine; Ketorolac; Loperamide; Metoclopramide; phenazepam; Benzodiazepines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Pregabalin (Experimental): This group (N= 40) receives up to 600 mg a day of Pregabalin for six-seven days along with symptomatic therapy that is divided into basic treatment that is given to all patients (Doxylamin 30 mg/day) and additional medications based on patients' needs as determined by a psychiatrist using the Opioid Withdrawal Scale and included Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine).
  Interventions: Drug: Pregabalin; Drug: Doxylamin; Drug: Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine)
- Clonidine (Active Comparator): This group (N= 40) receives up to 600 micrograms of Clonidine a day for six-seven days along with symptomatic therapy that is divided into basic treatment that is given to all patients (Doxylamin 30 mg/day) and additional medications based on patients' needs as determined by a psychiatrist using the Opioid Withdrawal Scale and included Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine)..
  Interventions: Drug: Clonidine; Drug: Doxylamin; Drug: Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine)

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 600 mg a day for six-seven days along with symptomatic therapy: Doxylamin 30 mg/day, Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine).
  Arms: Pregabalin
Drug: Clonidine — Clonidine 600 micrograms a day for six-seven days along with symptomatic therapy: Doxylamin 30 mg/day, Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine)
  Arms: Clonidine
Drug: Doxylamin
Drug: Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine)

SUMMARY:
It is a single blind randomized symptom triggered study to assess efficacy and safety of pregablin combined with the symptom triggered treatment for opiate withdrawal syndrome vs. clonidne with the same with the symptom triggered treatment for opiate withdrawal syndrome.

DETAILED DESCRIPTION:
Study design: Single-blind randomized symptom-regulated protocol with an active control. Eighty patients admitted to an inpatient addiction treatment program will be randomly assigned to two groups. The first group (N=40) receives up to 600 mg a day of Pregabalin for six days along with symptomatic therapy that is divided into basic treatment that is given to all patients (Doxylamin 30 mg/day) and additional medications based on patients' needs as determined by a psychiatrist using the Opioid Withdrawal Scale and included Ketorolac, Loperamide, Metoclopramide, Nefazolin and Phenazepam (benzodiazepine). The second group (N= 40) receives up to 600 micrograms of Clonidine a day as the main treatment along with the same basic and symptomatic regimen. Opiate withdrawal severity, craving, sleep disturbance, anxiety and depression, as well as general clinical impressions and side effects are assessed daily by psychiatrists who are blind to patients' group assignment using internationally validated quantitative psychometric instruments.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Use Disorders; Opioid Withdrawal Syndrome

Exclusion Criteria:

* Severe psychiatric and somatic disorders, other Substance Use Disorders (except tobacco)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of patients completed detoxification | 7 days
  Compares number of patients that finish treatment of opioid withdrawal syndrome (detoxification) in two treatment arms.

SECONDARY OUTCOMES:
Severity of opiod withdrawal | 7 days
  Compares changes of severity of opioid withdrawal syndrome in two arms
Amount of Ketorolac administered | 7 days
  Compares amount of Ketorolac administered under the symptom triggered protocol (per patient's request of physician's judgement) in two arms.
Number and severity of adverse events | 7 days
  Compares number and severity of adverse events in two treatment arms

OTHER OUTCOMES:
Craving for opiates | 7 days
  Craving for opiates will be measured with the visual analog scale. Compares craving for opiates in two treatment arms during detoxification.

CONTACTS AND LOCATIONS:
Locations (1):
- St.-Petersburg Bekhterev Reserach Psychoneurological Institute, Saint Petersburg, Russia